CLINICAL TRIAL: NCT00753285
Title: Renal Denervation in Patients With Refractory Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-040
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal Denervation (Experimental)
  Interventions: Device: Renal Denervation

INTERVENTIONS:
Device: Renal Denervation
  Other Names: Symplicity Renal Denervation System

SUMMARY:
The purpose of this study is to investigate the clinical utility of renal denervation for the treatment of refractory hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Systolic blood pressure of 160 mmHg or greater
* On 3 or more antihypertensive medications
* eGFR >= 45 mL/min

Exclusion Criteria:

* Renal artery abnormalities
* Known secondary hypertension attributable to a cause other than sleep apnea
* MI, angina, CVA within 6 months
* Type 1 diabetes
* Others

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Safety - complications associated with delivery and/or use of the Ardian Catheter, adverse renal events, electrolyte disturbances, hemodynamic events. | Through 3 years

SECONDARY OUTCOMES:
Physiologic response to renal denervation (e.g., blood pressure reduction) | Through 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, PhD, Principal Investigator — Monash University and the Alfred Hospital
Locations (3):
- United States (3):
  - Prairie Heart Institute, Springfield, Illinois
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - MetroHealth Medical Center, Cleveland, Ohio

REFERENCES:
- [Derived] Krum H, Schlaich MP, Sobotka PA, Bohm M, Mahfoud F, Rocha-Singh K, Katholi R, Esler MD. Percutaneous renal denervation in patients with treatment-resistant hypertension: final 3-year report of the Symplicity HTN-1 study. Lancet. 2014 Feb 15;383(9917):622-9. doi: 10.1016/S0140-6736(13)62192-3. Epub 2013 Nov 7. PMID 24210779
- See also: Medtronic Renal Denervation Program — http://www.medtronicrdn.com/index.htm